CLINICAL TRIAL: NCT04641403
Title: Laparoscopic-assisted Transversus Abdominis Plane Block for Post-laparoscopic Cholecystectomy Pain: A Prospective Double-blind Randomized Study '' .
Brief Title: "The Efficiency of Laparoscopic-assisted Transversus Abdominis Plane Block for Post-laparoscopic Cholecystectomy Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Private Medicabil Hospital (Other)
Responsible Party: Principal Investigator, Halil Özgüç, staff of general surgery, Private Medicabil Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MedicabilH
Record Dates: First submitted 2020-11-20; First posted 2020-11-23 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain
Keywords: Transversus abdominis plane block, postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: prospective randomized double blind
Who Masked: Participant, Care Provider
Masking Description: Anesthesia team, the patient, and the clinical nurses who carry out and record the postoperative evaluation will blinded to the group of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Standard IV analgesia group (SA), n=40): (No Intervention): In this group, the block will be administered with normal saline (NS) and all port sites will be infiltrated with NS.
- Group 2 (Local analgesia group (LA), n=40): (Active Comparator): In this group, the block wiil be administered with NS and local anesthetic will be administered to the port sites.
  Interventions: Procedure: The surgeon performed Laparoscopic-assisted TAP (LTAP) block
- Group 3 (two qudrant-Laparoscopic-assisted transversus abdominis plane block (LTAP) group, n=40) (Experimental): After the infiltration of all ports sites with NS, right sided two-quadrant block will be performed using bupivacaine.
  Interventions: Procedure: The surgeon performed Laparoscopic-assisted TAP (LTAP) block
- roup 4 (Four qudrant-Laparoscopic-assisted transversus abdominis plane block (LTAP) group, n=40) (Experimental): After the infiltration of all ports sites with NS, bilateral four-quadrant block will be performed using bupivacaine.
  Interventions: Procedure: The surgeon performed Laparoscopic-assisted TAP (LTAP) block

INTERVENTIONS:
Procedure: The surgeon performed Laparoscopic-assisted TAP (LTAP) block — After the induction of anesthesia, the first port will be inserted through the umbilicus and a 12 mmHg pneumoperitoneum will establish as a standard. Under the direct view of the laparoscopic camera, the block will be performed by inserting a 22-G needle just above the iliac crest through the midclavicular line posteriorly into the triangle of Petit and then inserting the needle below the costal arch through the midclavicular line towards the anterior axillary line into the subcostal plane. The block needle will be advanced under direct view until the two pops were felt and the extraperitoneal space will reach without puncturing the parietal peritoneum, and pulling back the needle 0.5 cm, the area of the thin transversus abdominis muscle fibers wiil be infiltrated. In this area, the correct plane of the needle tip will confirm by observing Doyle's bulge and the spread of the local anesthetic.
  Other Names: Standart İntravenous analgesia
  Arms: Group 2 (Local analgesia group (LA), n=40):; Group 3 (two qudrant-Laparoscopic-assisted transversus abdominis plane block (LTAP) group, n=40); roup 4 (Four qudrant-Laparoscopic-assisted transversus abdominis plane block (LTAP) group, n=40)

SUMMARY:
Laparoscopic cholecystectomy (LC) is a minimally invasive surgical procedure that causes moderate pain in the early postoperative period. In this prospective randomized study, the efficacy of four-quadrant and two-quadrant laparoscopic-assisted transversus abdominis plane (LTAP) block on postoperative pain will be compared with that of only intravenous analgesia (SA) and port-site infiltration of local anesthetic (LA).

Patients undergoing elective LC will be divided into four groups of 40 patients each using a randomization scale. The standard analgesia group will receive LTAP block with normal saline (NS) and port-site infiltration of NS, the LA group will receive LTAP block with NS and port-site infiltration of bupivacaine, while the four and two quadrant LTAP group will receive the block with bupivacaine and port-site infiltration of NS. Postoperative analgesia will be administered to all groups as a standard procedure. The patients' demographic data, postoperative 1, 3, 6, 12, and 24-hour visual analog pain (VAS) scores at rest and on cough, opioid requirement, presence of nausea and vomiting, and satisfaction scores will record in a standard form. The statistical analysis will be carried out using the SPSS software and the level of significance was set at p<0.05.

DETAILED DESCRIPTION:
This prospective, randomized, controlled, observer and patient-blind study will be conducted by the General Surgery, Anesthesiology and Reanimation Departments of Private Medicabil Hospital in accordance with the Declaration of Helsinki and Good Clinical Practice Guidelines. Hospital ethics committee approval was obtained for the study and the study was conducted between january 2021 and april 2020. Informed consent for the study to be conducted will obtained from each patient.

Study Inclusion and Exclusion Criteria The study will included American Society Anesthesia (ASA) 1 and 2 patients aged 18-70 years who underwent conventional four-quadrant LC.

Exclusion criteria:

1. Patients who did not agree to participate in the study,
2. ASA 3 and above patients, those who will undergone emergency surgery, open cholecystectomy
3. BMI of >40,
4. İntraoperative major complications,
5. History of severe allergy,
6. Chronic analgesic use, Study Parameters

1. gender, age, presence of comorbidity, weight, height, smoking status, operative time, length of hospital stay, intraoperative fluid volume, and developed complications 2. the primary data of the study: the postoperative 1, 3, 6, 12, and 24-hour VAS scores (0 lowest-10 highest) at rest and on cough after surgery 3. the rate of rescue analgesic dose of tramadol 4. as the secondary data: nausea-vomiting, shoulder pain, discharge duration exceeding 24 hours, and pre-discharge patient satisfaction (strongly disagree 1-strongly agree 5 on a Likert-type scale).

The mean postoperative 1-hour Visual Analog Scale (VAS) scores and the rates of rescue analgesic use of 20 patients operated before the study were determined. With these values, it was calculated that there should be 40 patients in each group, with a 33% decrease in pain scores and rescue analgesic use after LTAP at a statistical power of 80% and a significance level of 5%. The study was conducted with 30 patients in each group for a better analysis.

Randomization Randomization will be performed immediately before the surgery using a computer-generated random number table and was reported to the surgeon who would perform the surgery. Anesthesia team, the patient, and the clinical nurses who carry out and record the postoperative evaluation will blinded to the group of patients.

Procedure and Study Groups

The study groups were planned as follows:

Group 1 (Standard IV analgesia group (SA), n=40):

Group 2 (Local analgesia group (LA), n=40):

Group 4 (Four qudrant-Laparoscopic-assisted transversus abdominis plane block (LTAP) group, n=40) Postoperative analgesic administration will be carried out following a standard protocol in all groups. Acetaminophen 1 g was gradually will administered every 6 hours depending on the level of pain, and diclofenac sodium will intravenously administered every 12 hours depending on the requirement. In the case of a pain score above 4, tramadol 100 mg will be given intravenously as a rescue analgesic.

Block technique:

After the induction of anesthesia, the first port was inserted through the umbilicus and a 12 mmHg pneumoperitoneum was established as a standard. Under the direct view of the laparoscopic camera, the block was performed by inserting a 22-G needle just above the iliac crest through the midclavicular line posteriorly into the triangle of Petit and then inserting the needle below the costal arch through the midclavicular line towards the anterior axillary line into the subcostal plane. The block needle was advanced under direct view until the two pops were felt and the extraperitoneal space was reached without puncturing the parietal peritoneum, and pulling back the needle 0.5 cm, the area of the thin transversus abdominis muscle fibers was infiltrated. In this area, the correct plane of the needle tip was confirmed by observing Doyle's bulge and the spread of the local anesthetic.11,14 This procedure was performed as the bilateral four-quadrant block in BLTAP group and right sided two-quadrant block in ULTAP group.

Statistical Analysis The SPSS (IBM SPSS, version20) software will be used for the statistical analysis. The t-test was will use for continuous variables, while the chi-square test for categorical values. The level of significance was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesia (ASA) 1 and 2 patients aged 18-70 years

Exclusion Criteria:

* 1. Patients who did not agree to participate in the study, 2. ASA 3 and above patients, those who will undergone emergency surgery, open cholecystectomy 3. BMI of >40, 4. İntraoperative major complications, 5. History of severe allergy, 6. Chronic analgesic use,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain score | postoperatively 1,3,6,12 and 24 hours
  he postoperative 1, 3, 6, 12, and 24-hour VAS scores (0 lowest-10 highest) at rest and on cough after surgery

SECONDARY OUTCOMES:
satisfaction score | postoperatively 24 hours
  nausea-vomiting, shoulder pain, discharge duration exceeding 24 hours, and pre-discharge patient satisfaction (strongly disagree 1-strongly agree 5 on a Likert-type scale).

CONTACTS AND LOCATIONS:
Overall Officials: Halil Özgüç, md, Principal Investigator — Medical Doctor
Locations (1):
- Private Medicabil Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cevikkalp E, Narmanli M, Ozguc H, Ocakoglu G. Bilateral 4-quadrant laparoscopic-assisted transversus abdominis plane block reduces early postoperative pain after laparoscopic cholecystectomy: A prospective, single-blind, randomized study. Saudi Med J. 2023 Feb;44(2):145-154. doi: 10.15537/smj.2023.44.2.20220407. PMID 36773971